CLINICAL TRIAL: NCT06438861
Title: Exploring the Additive Effect of Vibegron to Intradetrusor OnabotulinumtoxinA in Women With Refractory Overactive Bladder
Brief Title: Role of Combination Therapy in Women With Refractory Overactive Bladder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded by industry
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Katelyn Donaldson, MD, Urogynecology Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300012698; Pending (Other Grant/Funding Number: Pending)
Record Dates: First submitted 2024-05-15; First posted 2024-06-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Overactive Bladder Syndrome
Keywords: Refractory Overactive Bladder Syndrome
MeSH Terms: interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 100U intradetrusor onabotulinumtoxinA plus vibegron (Active Comparator): Each patient will undergo intradetrusor onabotulinumtoxinA injections of 100U either in the office or in the operating room depending on patient and provider preference. Patients randomized to this arm will begin taking vibegron 75mg daily, which is the standard dose, starting the day of their procedure and continue for 3 months.
  Interventions: Drug: Vibegron 75mg
- 100U intradetrusor onabotulinumtoxinA plus placebo (Placebo Comparator): Each patient will undergo intradetrusor onabotulinumtoxinA injections of 100U either in the office or in the operating room depending on patient and provider preference. Patients randomized to this arm will begin taking a placebo pill daily starting the day of their procedure and continue for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vibegron 75mg — Each patient will undergo intradetrusor onabotulinumtoxinA injections of 100U either in the office or in the operating room depending on patient and provider preference. Patients will begin taking vibegron 75mg daily or a placebo pill daily starting the day of their procedure and continue for 3 months.
  Arms: 100U intradetrusor onabotulinumtoxinA plus vibegron
Drug: Placebo — Each patient will undergo intradetrusor onabotulinumtoxinA injections of 100U either in the office or in the operating room depending on patient and provider preference. Patients will begin taking vibegron 75mg daily or a placebo pill daily starting the day of their procedure and continue for 3 months.
  Arms: 100U intradetrusor onabotulinumtoxinA plus placebo

SUMMARY:
Defined by the International Continence Society (ICS) as urinary "urgency, with or without urge incontinence, usually with frequency and nocturia", overactive bladder (OAB) presents as challenging syndrome to treat. OAB is a very prevalent condition, affecting between 11.8% to 16% of the population with equal impact on women and men and growing prevalence with age. OAB is associated with a significant financial burden to both patients and the health care system with a estimated cost of US $82.6 billion in 2020. Traditionally, a stepwise approach has been taken in managing OAB; starting first with lifestyle modifications, followed by anticholinergic or beta-3-agonist medications as the second line, and lastly, intradetrusor onabotulinumtoxinA injections, percutaneous tibial nerve stimulation (PTNS), and sacral neuromodulation (SNM) as third line options. Given the limitations of this stepwise approach in patients with refractory OAB, combination therapy offers patients an increasing number of treatment options but the literature surrounding the efficacy of combination therapy is somewhat limited. A 2019 systematic review revealed there were only 32 studies in the current OAB literature that explored the role of combination therapy, and the majority of these studies examined the effect of lifestyle modifications with another intervention strategy, highlighting an untapped area of research5.

To date, there has only been a single pilot study conducted in Taiwan examining the effect of intradetrusor onabotulinumtoxinA injections with the addition of mirabegron for patients with refractory OAB. This study by Wang et al. explored the therapeutic impact of adding either an anticholinergic, solifenacin, or a beta-3 agonist, mirabegron, to intradetrusor onabotulinumtoxinA injections as compared to each other as well as patients receiving onabotulinumtoxinA alone. Ninety patients were enrolled with 30 patients allocated to the solifenacin arm, 31 to the mirabegron arm, and 29 to the control group. While the baseline data among the three arms was comparable, the percentage of OAB wet in the mirabegron plus onabotulinumtoxinA group was significantly less at 3-, 6-, 9-, and 12-month intervals than the solifenacin plus onabotulinumtoxinA and the onabotulinumtoxinA alone groups. While this pilot study reveals the potential additive benefit of a beta-3 agonist to intradetrusor onabotulinumtoxinA, no further studies have been performed to date and there are no studies regarding the additive benefit of vibegron, which has a more tolerable side effect profile and is not as limited by as many contraindications as mirabegron. If vibegron can potentiate the effect of intradetrusor onabotulinumtoxinA, this presents a new treatment strategy for OAB and could offer patients an additional line of therapy before having to pursue more invasive and costly management option of sacral neuro modulation.

DETAILED DESCRIPTION:
The study will be a prospective double-blinded randomized control trial to examine the effect of administering vibegron versus placebo in conjunction with intradetrusor onabotulinumtoxinA injections for the management of refractory OAB. Patients who present to the University of Alabama at Birmingham urogynecology practice with refractory OAB undergoing the standard 100U intradetrusor onabotulinumtoxinA will be offered enrollment to either the onabotulinumtoxinA plus vibegron or the onabotulinumtoxinA plus placebo groups. Prior to onabotulinumtoxinA injections, patients' baseline demographics will be documented and their genitourinary symptoms will be assessed using the previously validated Urinary Distress Inventory Short Form (UDI-6), the Incontinence Impact Questionnaire Short Form (IIQ-7), the Overactive Bladder Questionnaire (The OAB-q), and a 3 day voiding diary. Patients will be blinded to which cohort they are randomized to. Each patient will undergo intradetrusor onabotulinumtoxinA injections of 100U either in the office or in the operating room depending on patient and provider preference. Patients will begin taking vibegron or a placebo pill daily starting the day of their procedure. At 12 weeks, patients will complete a 3 day voiding diary as well as the UDI-6, IIQ-7, and OAB-q questionnaires. Patient charts will be queried for timing of repeat onabotulinumtoxinA injection as another secondary outcome.

Primary outcome: Change in mean urinary urgency incontinence episodes at 12 weeks based on 3 day voiding diary

Secondary outcomes: Mean change in UDI-6 responses at 12 weeks, mean change in IIQ-7 responses at 12 weeks, mean change in OAB-q responses at 12 weeks, duration to repeat onabotulinumtoxinA injection

Sample Size Calculation:

It is anticipated that women randomized to the 100U intradetrusor onabotulinumtoxinA plus vibegron arm will experience a greater improvement in UUI episodes compared to the 100U intradetrusor onabotulinumtoxinA plus placebo cohort. A recent study comparing the PTNS plus mirabegron to PTNS plus placebo performed a sample size calculation using existing data 7,8. In that calculation, a 2-sided alpha=0.05, the estimate for that difference in improvement had been estimated to be 2.5 UUI episodes over a 3-day bladder diary pre-vs. post-treatment with a standard deviation of 3 and a power of 0.80 and given the assumed attrition rate of 10%, the total N per arm was estimated to be 27 subjects for the study. Given the similarities between this study and our proposed study, the sample size calculation was felt be applicable to this study.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing intradetrusor botulinum injections for refractory OAB
2. Age 18 years old or greater
3. Fluency and literacy in English
4. Capacity to provide consent

Exclusion Criteria:

1. Allergy to Vibegron
2. Currently pregnant or planning to become pregnant
3. Breastfeeding
4. Current digoxin use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in urinary urgency incontinence (UUI) episodes on 3 day voiding diary at 12 weeks after starting treatment as compared to baseline | Pre-intervention baseline to 12 weeks following initiation of intervention
  Patients will be asked to complete a 3 day voiding diary at baseline and at 12 weeks following intradetrusor onabotulinumtoxinA injections and oral medication. The mean change in UUI episodes will be compared between the onabotulinumtoxinA injection plus vibegron verus onabotulinumtoxinA injection plus placebo groups.

SECONDARY OUTCOMES:
Change in Symptom Distress as Measured by the Urogenital Distress Index (UDI-6) Questionnaire Pre-Intervention versus 12 weeks Post-Intervention | Pre-intervention baseline to 12 weeks following initiation of intervention
  The UDI-6 is the short form validated patient questionnaire that was developed from the urogenital distress inventory (UDI). It consists of six questions that focus on lower urinary tract dysfunction including obstructive, irritative, and stress symptoms. The responses are scored as follows: (0) not at all, (1) slightly, (2) moderately, (3) greatly. The mean score is multiplied by 33 1/3 to convert to a 0 to 100 scale with higher scores indicative of more symptoms distress. Subjects will complete the UDI-6 survey at baseline and at 12 weeks post-intervention. The mean change in UDI-6 responses will be compared.
Change in UUI (Urge Urinary Incontinence)/OAB (Overactive Bladder) Quality of Life as Measured by the Incontinence Impact Questionnaire Short Form (IIQ-7) Questionnaire Pre-Intervention versus 12 weeks Post-Intervention | Pre-intervention baseline to 12 weeks following initiation of intervention
  The IIQ-7 is the short form validated patient questionnaire that was developed from the incontinence impact questionnaire (IIQ). It consists of seven questions that focus on the impact of UUI on physical activity, travel, relationships, and emotional health. The responses are scored as follows: (0) not at all, (1) slightly, (2) moderately, (3) greatly. The mean score is multiplied by 33 1/3 to convert to a 0 to 100 scale with higher scores indicative of more symptoms distress. Subjects will complete the IIQ-7 survey at baseline and at 12 weeks post-intervention. The mean change in IIQ-7 responses will be compared.
hange in UUI (Urge Urinary Incontinence)/OAB (Overactive Bladder) Quality of Life as Measured by the Overactive Bladder Questionnaire-Short Form (OAB-q SF) Questionnaire Pre-Intervention versus 12 weeks Post-Intervention | Pre-intervention baseline to 12 weeks following initiation of intervention
  The OAB-q SF is the short form validated patient questionnaire that was developed from the Overactive Bladder Questionnaire (OAB-q). It consists of six questions that focus on the impact of bladder symptoms over the past 4 weeks. The responses are scored as follows: (1) not at all, (2) a little bit, (3) somewhat, (4) quite a bit, (5) a great deal, (6) a very great deal. The mean score is converted to a 0 to 100 scale with higher scores indicative of more symptoms distress. Subjects will complete the OAB-q SF survey at baseline and at 12 weeks post-intervention. The mean change in OAB-q SF responses will be compared.
Duration to repeat onabotulinumtoxinA injection | Initiation of intervention until repeat injection, anticipate average of 1 year
  Patient require repeat intradetrusor onabotulinumtoxinA injection to treat refractory OAB. A chart review will be performed to determine time interval between initial onabotulinumtoxinA injection and subsequent injection to see if there is a difference with the addition of vibegron as compared to placebo.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Coyne KS, Wein A, Nicholson S, Kvasz M, Chen CI, Milsom I. Economic burden of urgency urinary incontinence in the United States: a systematic review. J Manag Care Pharm. 2014 Feb;20(2):130-40. doi: 10.18553/jmcp.2014.20.2.130. PMID 24456314
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Kasman A, Stave C, Elliott CS. Combination therapy in overactive bladder-untapped research opportunities: A systematic review of the literature. Neurourol Urodyn. 2019 Nov;38(8):2083-2092. doi: 10.1002/nau.24158. Epub 2019 Sep 4. PMID 31483070
- [Background] Wang CC, Lee CL, Hwang YT, Kuo HC. Adding mirabegron after intravesical onabotulinumtoxinA injection improves therapeutic effects in patients with refractory overactive bladder. Low Urin Tract Symptoms. 2021 Oct;13(4):440-447. doi: 10.1111/luts.12384. Epub 2021 May 6. PMID 33960119
- [Background] Sancaktar M, Ceyhan ST, Akyol I, Muhcu M, Alanbay I, Mutlu Ercan C, Atay V. The outcome of adding peripheral neuromodulation (Stoller afferent neuro-stimulation) to anti-muscarinic therapy in women with severe overactive bladder. Gynecol Endocrinol. 2010 Oct;26(10):729-32. doi: 10.3109/09513591003649815. PMID 20210697
- [Background] Stanley RF, Meyer I, Blanchard CT, Richter HE. Posterior Tibial Nerve Stimulation With versus Without Mirabegron: A Randomized Controlled Trial. Int Urogynecol J. 2024 Aug;35(8):1709-1717. doi: 10.1007/s00192-024-05835-y. Epub 2024 Aug 5. PMID 39101958